CLINICAL TRIAL: NCT07141017
Title: Evaluating the Impact of an Initial Standardized Global Review in Patients With Early Axial Spondyloarthritis: a Multicenter Randomized Cluster-controlled Study
Brief Title: Initial Standardized Global Review in Axial Spondyloarthritis
Acronym: REVINSPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Recherche Clinique en Rhumatologie (Other)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A02314-43
Record Dates: First submitted 2025-07-29; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Axial Spondylarthritis (axSpA)
Keywords: Rheumatology; Initial standardized global review

STUDY DESIGN:
Intervention Model Description: The study will be a cluster-randomized, controlled study with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Other: Initial standardized global review
- Usual care arm (No Intervention)

INTERVENTIONS:
Other: Initial standardized global review — The intervention under study will be the initial standardized global review, which will be performed as soon as axial spondyloarthritis is diagnosed (less than 12 months from diagnosis is mandatory) and only at the baseline visit.
  This review includes both the assessment of different domains of the disease, but also the education and information on such different domains of the disease and its management
  The domains assessed during the intervention will be: diagnosis of spondyloarthritis, spondyloarthritis phenotype, disease activity, disease severity and function, treatment adherence and comorbidities.
  At the end of the intervention, a detailed medical report on this initial standardized global review will be produced and sent to the patient, their rheumatologist, their general practitioner, and their dispensing pharmacist.
  Arms: Intervention arm

SUMMARY:
This study will be a pragmatic, cluster-randomized, controlled study with two parallel arms ( 'intervention' and 'usual care' (UC) arms) of one year duration.

The study will be open-label, but centers randomized in the UC arm will not be aware of the intervention performed in the 'intervention' centers.

The primary objective of this study will be to determine whether participation in a standardized global review (that includes assessment of disease domains and education ) as soon as possible after diagnosis of axial spondyloarthritis has a beneficial impact on patient knowledge of the disease at 12 months. The primary endpoint will be the change in the SPAKE (SPondyloArthritis Knowledge Questionnaire) questionnaire between M0 and M12.

ELIGIBILITY:
Inclusion Criteria:

* Adults (but age <80years) with a diagnosis of axial spondyloarthritis determined by the treating rheumatologist within the 12 months preceding the baseline visit, who have completed the informed consent and have the ability to complete all study activities.

Exclusion Criteria:

* Patients who have already received a specific (or plan to receive in the coming 12 months) and dedicated program/global evaluation including education on the disease or treatments.
* Patients with any physical or mental condition that may affect understanding of the intervention or adherence to treatment (e.g. major depression or substance/alcohol use - might have impact on the outcomes of interest in the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The change in patient knowledge of the disease. | Visits Day 0 and Month 12
  The primary endpoint will be the change in the SPAKE questionnaire

SECONDARY OUTCOMES:
Treatment | Visits Day 0 and Month 12
  Treatment in both groups will be evaluated NSAID intake and % of patients receiving csDMARD/bDMARD/tsDMARD
The ability to cope with the disease | Visits Day 0 and Month 12
  The ability to cope with the disease will be evaluated by disease coping change between Day 0 and Month 12 in both groups using the Coping Scale from the RAID questionnaire
Knowledge on b/tsDMARDs | Visits Day 0 and Month 12
  Knowledge on b/tsDMARDs, only in patients with b/tsDMARD, will be evaluated by the BioSECURE'21 questionnaire
Adherence to axSpA treatments | Visits Day 0 and Month 12
  Adherence to axSpA treatments in both groups will be evaluated by the CQR5 questionnaire
Disease activity | Visits Day 0 and Month 12
  Disease activity will be evaluated by the disease activity score (ASDAS) change in both groups
Number of comorbidities | Visit Month 12
  Number of comorbidities managed according to recommendations in both groups
Function change | Visits Day 0 and Month 12
  Function change in both groups between will be evaluated by the BASFI questionnaire
Quality of life change | Visits Day 0 and Month 12
  Quality of life change in both groups will be evaluated by the ASAS-HI questionnaire
Work impairment | Visit Month 12
  Work impairment will be evaluated by the WPAI questionnaire
Assessment of health services resources use | Visit Month 12
  Assessment of health services resources use will be evaluated by self-questionnaire
The patient's perception of the benefits of this type of initial global standardized review on patient's follow-up and the treating rheumatologist's perception of the benefits of this type of initial global standardized review on patient follow-up | Visit Month 12
  The patient's perception of the benefits of this type of initial global standardized review on patient's follow-up and the treating rheumatologist's perception of the benefits of this type of initial global standardized review on patient follow-up will be evaluated by the Likert scale
The sources of information accessed by patients | Visits Day 0 and Month 12
  The sources of information accessed by patients in both groups be evaluated with the percentage of patients who participated in a therapeutic education programme

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHRU Brest - Hôpital de La Cavale Blanche, Brest
  - CHU Caen, Caen
  - CHU Clermont-Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - AP-HP - Hôpital Henri Mondor, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - AP-HP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - GHICL - Hôpital Saint Philibert, Lomme
  - AP-HM - Hôpital St Marguerite, Marseille
  - AP-HP - Hôpital Cochin, Paris
  - AP-HP - Hôpital La Pitié Salpétrière, Paris
  - AP-HP - Hôpital Lariboisière, Paris
  - AP-HP - Hôpital Saint Antoine, Paris
  - HCL - Hôpital Lyon Sud, Pierre-Bénite
  - CHU Rouen - Hôpital Charles-Nicolle, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Hopitaux de Toulouse (CHU) - Hôpital Pierre Paul Riquet, Toulouse
  - CHU Tours - Hôpital Trousseau, Tours